CLINICAL TRIAL: NCT04762316
Title: Uterine Fibroids Are a Prevalent Finding in Women of Reproductive Age. Ready Safety Study Extracts of Plants Pregnenolone, Pyridoxal Phosphate, and Dydrogesterone for Treating Uterine Fibroids in Women's Pregnancy.
Brief Title: Composition for Treating Uterine Fibroid (SB-UF)
Acronym: SB-UF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Trieu, Nguyen Thi, M.D. (Individual)
Collaborators: TRAN MINH DUC, MD (Unknown); Tran Minh Cam Tu, MD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Removal the Uterine Fibroids
Record Dates: First submitted 2021-01-03; First posted 2021-02-21 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Uterine Fibroids Affecting Pregnancy
MeSH Terms: interventions — Pregnenolone; Pyridoxal Phosphate; Dydrogesterone

STUDY DESIGN:
Intervention Model Description: Selection of women ages 18 to 40, with pregnancy uterine fibroids and pregnancy in the 8th week of pregnancy.
Who Masked: Participant, Investigator
Masking Description: The number of post-recruiting people who have fibroids is divided into 2 groups
  * The group of pregnancy uterine fibroids uses drugs under study.
  * The group of pregnancy uterine fibroids uses a placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SB-UF Drug (Experimental): Use SB-UF drugs to lose the size of Uterine Fibroids on Women the Pregnancy. Measuring the size of uterine fibroid. Monitor the disappearance of uterine fibroids from 4 - 40 weeks
  Interventions: Drug: SB-UF
- SB-UF Placebo (Placebo Comparator): Use SB-UF placebo to lose the size of Uterine Fibroids on Women the Pregnancy. Measuring the size of uterine fibroid. Monitor the disappearance of uterine fibroids from 4 - 40 weeks
  Interventions: Device: SB-UF Placebo

INTERVENTIONS:
Drug: SB-UF — Dosage:
  -Take 1tablet/2 times/day/in throughout pregnancy.
  Other Names: Pregnenolone 60mg & Pyridoxal Phosphate 20mg & Dydrogesterone 10mg & Impatien balsamina extract 100 mg
  Arms: SB-UF Drug
Device: SB-UF Placebo — Dosage:
  -Take 1tablet/2 times/day/in throughout pregnancy.
  Other Names: Pregnenolone & Pyridoxal Phosphate Placebo
  Arms: SB-UF Placebo

SUMMARY:
Pregnenolone & Pyridoxal Phosphate SB-UF for treating uterine fibroids in women's pregnancies to lose the size of fibroids and to dissolve fibroids.

Uterine fibroids are a very common finding in women pregnancy of reproductive age, fibroids fast grow in the first trimester of pregnancy. SB-UF against the rapid growth of fibroids under the influence of hormones during pregnancy. Use SB-UF to think about regulating stable Oestrogen levels and dissolving fibroids.

This is a substantial insight into disease pathogenesis, with a clear path toward clinical application, which would lead to a substantial advance and perfection in management or public health policy.

DETAILED DESCRIPTION:
Uterine fibroids are a very common finding in women's pregnancy of reproductive age fibroids fast grow in the first trimester of pregnancy.

Clinically has shown that:

* Uterine fibroids are associated with heavy or prolonged menstrual periods, and abnormal bleeding between menstrual periods.
* Fibroids are associated with increased rates of spontaneous miscarriage, premature birth, placenta ablation, malpresentation, labor dysfunction, cesarean section, and postpartum hemorrhage, pain is the most common complication of fibroids uterus during pregnancy.
* Use the composition that has sufficient Pregnenolone, and coenzyme Pyridoxal Phosphate, and combined with Dydrogesterone, this preparation will soften uterine fibroids and disappear fibroids.

Pregnenolone is produced in the adrenal glands and the central nervous system. Pregnenolone is synthesized from Cholesterol and it is the precursor of Progesterone, Estrogen, and dehydroepiandrosterone (DHEA). In some people Pregnenolone will decrease with age, which will lead to an imbalance between Progesterone and estrogen, according to research, this imbalance is the cause of abnormal growth of the uterine muscle fibers cells that produce multiple fibroids in the womb. Supplementation Pregnenolone is necessary for women of childbearing and reproductive age, overtime tracking pregnant women but there were fibroids from before pregnancy these fibroids will develop very quickly to stun the fetus many problems in pregnancy, and childbirth, the risk of miscarriage, preterm delivery,...The new drug will maintain a sufficient amount of Pregnenolone natural is the essence from Dioscorea persimilis prain & burkill and associated with a necessary element is Coenzyme Pyridoxal Phosphate, Dydrogesterone. Compound presence in the body will curb the development of the muscle fibers uterus, the muscle fibers in the fibroids will soften, spread out, and disappear fibroids. The uterus returns to its normal state, the fetus will develop naturally.

Research results

* After 40 weeks of ultrasound examination:

  * 100% of women using SB-UF drugs have the disappearance of fibroids, only the image of uterine muscle is thicker than usual.
  * 100% of women who received SB-UF placebo did not experience any beneficial progress.
* Through study completion, an average of 40 weeks

ELIGIBILITY:
Inclusion Criteria:

* Procedure to the treatment of fibroids in pregnancy and in women desiring future fertility.

Exclusion Criteria:

* Subserosal fibroids may be pedunculated hanging from a stalk inside or outside the uterus.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women aged 18 to 40 years who are pregnant and have uterine fibroids in the following forms: Intramural fibroids, Submucosal fibroids, Subserous fibroids.
Enrollment: 66 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Use SB-UF drugs to lose the size of Uterine Fibroids on Women the Pregnancy. | 40 weeks
  Measuring the size of uterine fibroid. Monitor the disappearance of benign smooth muscle cell tumors of the uterus

CONTACTS AND LOCATIONS:
Overall Officials: Thi Trieu Nguyen, Dr., Principal Investigator — Trieu, Nguyen Thi, M.D.
Locations (2):
- Saigon Biopharma LLC, Wilmington, Delaware, United States
- Saigon Biopharma Company Limited, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Contemporary Management of Fibroids in Pregnancy — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2876319
- See also: Uterine fibroids — http://www.mayoclinic.org/diseases-conditions/uterine-fibroids/symptoms-causes/syc-20354288
- See also: WO2020095085 - COMPOSITION for TREATING UTERINE FIBROIDS — http://patentscope.wipo.int/search/en/detail.jsf?docId=WO2020095085&_cid=P20-KJGXFA-35465-1